CLINICAL TRIAL: NCT04646135
Title: Not for Profit, Monocentric, Open Label Trial of Lorazepam, Randomized to Three Different Sequences of Boli and Continuous Infusion, for Sedation of Children Aged ≥1 and <12 Years Admitted in Intensive Care and Mechanically Ventilated.
Brief Title: Lorazepam for the Analgosedation of Pediatric Patients in Mechanical Ventilation.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Collaborators: Ministero della Salute, Italy (Other); University College, London (Other)
Responsible Party: Principal Investigator, Marco Marano, Principal Investigator, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1954 / 2019; 2019-003901-93 (EudraCT Number)
Record Dates: First submitted 2020-06-18; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Analgesia
Keywords: Lorazepam; Intensive Care; Analgosedation; Mechanical Ventilation; Propylene Glycol
MeSH Terms: conditions — Agnosia | interventions — Lorazepam

STUDY DESIGN:
Intervention Model Description: Arm I:
  * Day 1: 6 Boluses at 0.1 mg/kg LZ every 4 hr
  * Day 2: 6 Boluses at 0.2 mg/kg LZ every 4 hr
  * Day 3: Continuous Infusion at 0.025 mg/kg/hr LZ
  Arm II:
  * Day 1: 6 Boluses at 0.2 mg/kg LZ every 4 hr
  * Day 2: 6 Boluses at 0.1 mg/kg LZ every 4 hr
  * Day 3: Continuous Infusion at 0.03 mg/kg/hr LZ
  Arm III:
  * Day 1: 6 Boluses at 0.3 mg/kg LZ every 4 hr
  * Day 2: 6 Boluses at 0.1 mg/kg LZ every 4 hr
  * Day 3: Continuous Infusion at 0.025 mg/kg/hr LZ
  Patients will be monitored for further 3 days of follow-up, after the end of the administration sequence. In case they would still need to undergo analgosedation, other drugs will be administered (e.g. midazolam, dexmedetomidine).
  Patients will also be divided into two age groups - 6 patients: age ≥1 year <5 years (COHORT 1); 3 patients: age ≥5 years - <12 years (COHORT 2)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sequence 1 (Experimental): The subjects enrolled in this arm, will undergo the following lorazepam administration scheme:
  * Day 1: 6 Boluses at 0.1 mg/kg LZ every 4 hours
  * Day 2: 6 Boluses at 0.2 mg/kg LZ every 4 hours
  * Day 3: Continuous Infusion at 0.025 mg/kg/hour LZ
  Interventions: Drug: Lorazepam 4 mg/ml
- Sequence 2 (Experimental): The subjects enrolled in this arm, will undergo the following lorazepam administration scheme:
  * Day 1: 6 Boluses at 0.2 mg/kg LZ every 4 hours
  * Day 2: 6 Boluses at 0.1 mg/kg LZ every 4 hours
  * Day 3: Continuous Infusion at 0.03 mg/kg/hour LZ
  Interventions: Drug: Lorazepam 4 mg/ml
- Sequence 3 (Experimental): The subjects enrolled in this arm, will undergo the following lorazepam administration scheme:
  * Day 1: 6 Boluses at 0.3 mg/kg LZ every 4 hours
  * Day 2: 6 Boluses at 0.1 mg/kg LZ every 4 hours
  * Day 3: Continuous Infusion at 0.025 mg/kg/hour LZ
  Interventions: Drug: Lorazepam 4 mg/ml

INTERVENTIONS:
Drug: Lorazepam 4 mg/ml — Lorazepam will be administered intravenously according to the scheduled sequences.

SUMMARY:
The aim of this study is to better define the pharmacokinetic and pharmacodynamic profile of lorazepam for the analgosedation in pediatric intensive care unit. This will help to better define the dosages and administration modalities (bolus or continue infusion) required to achieve analgosedation with lorazepam in pediatric patients undergoing mechanical ventilation.

DETAILED DESCRIPTION:
The prolonged use of certain sedative drugs such as midazolam, whose metabolism is associated with the production of active metabolites, can lead to difficult management of sedative therapy and ventilatory weaning. The active metabolites, whose production is variable, determine in fact a difficulty in establishing a precision therapy, thus making it necessary to identify new molecules for sedation in pediatric intensive care unit (PICU). Lorazepam (LZ) is a benzodiazepine with an intermediate duration of activity, administered by continuous infusion or intermittent bolus, which has the advantages of higher potency compared to other benzodiazepines, a low cost and a metabolism that does not produce active metabolites. However, the presence of propylene glycol (PG), an excipient present in intravenous LZ formulations, although generally well tolerated, is potentially associated with episodes of tissue toxicity due to accumulation phenomena; this may represent a risk in cases where LZ is administered in high doses. This study, based on pharmacokinetic models obtained from data already available in the scientific literature, aims to define the pharmacokinetic and pharmacodynamic characteristics of LZ for the analgosedation of pediatric patients admitted to intensive care and subjected to mechanical ventilation. Preliminary evaluation of sedative efficacy will be carried out through COMFORT-B scale assessment.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent of the parents or legal representatives of minors according to national law;
* Male and/or female subjects of the following ages: ≥1 year - <12 years;
* Critical patients who need to undergo mechanical ventilation and hospitalized in PICU;

Exclusion Criteria:

* Hospitalization in PICU expected to be less than 48 hours long;
* Altered renal function (eGFR according to Schwartz < 30 mL/min/1.73 m2 or creatininemia > 2 vn);
* Altered liver function (bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 2 NU);
* Altered cardiac function (Ejection Fraction < 50%);
* Need for administration of neuromuscular blocking drugs;
* Concomitant therapy with continuous infusion drugs containing PG;
* Metronidazole therapy in the three months prior to enrollment;
* History of exposure to LZ in the seven days prior to enrollment;
* Participation in other experimental clinical trials;
* Patient undergoing extracorporeal circulation (dialysis, ECMO)
* Known allergic reaction to LZ or its excipients;
* Weight < 9 kg;
* Known immaturity of the enzymatic system of alcohol dehydrogenase;
* Pregnancy in progress;
* Ingestion of antifreeze;
* Treatment with silver sulfadiazine for wound care;
* Oncological pathology diagnosed or suspected;
* Valproic acid therapy
* Patients undergoing continuous infusion therapy with drugs used for sedation prior to admission to the red area (excluding dexmedetomidine).

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Lorazepam Pharmacokinetics (AUC) | 72 hours from enrollment
  AUC of Lorazepam

SECONDARY OUTCOMES:
Analgosedative efficacy of Lorazepam | 72 hours from enrollment
  Frequency of responder patients (COMFORT-B scale score between 11 and 22 and alertness score between 2 and 3)
COMFORT-BEHAVIOURAL (COMFORT-B) scale | 72 hours from enrollment
  Median (IQR) of COMFORT-B scale score and alertness score. The COMFORT BEHAVIOURAL (COMFORT-B) SCALE consists of six items: alertness, calmness, respiratory response (for children undergoing mechanical ventilation), body movements, facial tension and muscle tone. Each item goes from 1 to 5, assessing the different intensities. The sum of the six ratings leads to a final score ranging from a minimum of 6 to a maximum of 30. A patient is considered to be under-sedated in case of COMFORT-B scores of 23 or higher, over-sedated in case of COMFORT-B scores of 10 or lower.
Dropouts due to any adverse event | 72 hours from enrollment
  Number of interruptions of the experimental administration sequence due to adverse events
Adverse Events (AEs)/ Serious Adverse Events (SAEs) registration at end of study | 72 hours from enrollment
  Number of AEs / SAEs at the end of the administration of the experimental drug
AEs/SAEs registration at end of follow-up | 6 days from enrollment
  Number of AEs / SAEs at the end of the follow-up period
Vital signs at the end of study (Blood Pressure) | 72 hours from enrollment
  Blood Pressure measurement in mmHg, change from baseline (Median (IQR))
Vital signs at the end of study (Heart Rate) | 72 hours from enrollment
  Heart rate measurement in beats per minute (b.p.m), change from baseline (Median (IQR))
Vital signs at the end of study (Body Temperature) | 72 hours from enrollment
  Body temperature measurement in °C, change from baseline (Median (IQR))
Vital signs at the end of follow-up (Blood Pressure) | 6 days from enrollment
  Blood Pressure measurement in mmHg, change from baseline (Median (IQR))
Vital signs at the end of follow-up (Heart Rate) | 6 days from enrollment
  Heart rate measurement in beats per minute (b.p.m), change from baseline (Median (IQR))
Vital signs at the end of follow-up (Body Temperature) | 6 days from enrollment
  Body temperature measurement in °C, change from baseline (Median (IQR))
Plasma concentrations of Propylene Glycol at the end of study | 72 hours from enrollment
  AUC of PG in mg/L in serum
Osmol gap at the end of study | 72 hours from enrollment
  Osmol gap (detected osmolarity - calculated osmolarity) change from baseline (Median (IQR)
C-Cystatin at the end of study | 72 hours from enrollment
  Plasma levels (AUC) of the early marker of kidney damage (C-Cystatin) changes from baseline
N-GAL at the end of study | 72 hours from enrollment
  Plasma levels (AUC) of the early marker of kidney damage (N-GAL) changes from baseline
Kidney Function at the end of study | 72 hours from enrollment
  Estimated Glomerular Filtration Rate (eGFR) change from baseline (Median (IQR))
Lorazepam Pharmacokinetics (Cmax) | 72 hours from enrollment
  Cmax of Lorazepam
Lorazepam Pharmacokinetics (Tmax) | 72 hours from enrollment
  Tmax of Lorazepam
Lorazepam Pharmacokinetics (Drug Clearance) | 72 hours from enrollment
  Drug clearance (CL)
Lorazepam Pharmacokinetics (Half Life) | 72 hours from enrollment
  Half life (t1/2) of Lorazepam
Lorazepam Pharmacokinetics (Cmin) | 72 hours from enrollment
  Cmin of Lorazepam

CONTACTS AND LOCATIONS:
Overall Officials: Marco Marano, MD, Principal Investigator — Bambino Gesù Hospital and Research Institute

IPD SHARING:
Plan to Share IPD: No